CLINICAL TRIAL: NCT07099690
Title: Perineal Massage During Labor for the Prevention of Perineal Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Gabriela Plentz Stein, Researcher, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-0514
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Obstetric; Injury Pelvic Floor
Keywords: Perineal trauma; Episiotomy; Perineal massage; Laceration
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineal Massage Group (Experimental): The perineal massage group will receive the intervention during labor.
  Interventions: Procedure: Perineal massage
- Control Group (No Intervention): The control group will receive the standard care provided by the obstetric center.

INTERVENTIONS:
Procedure: Perineal massage — Perineal massage will be performed during labor, either between or during contractions, regardless of the position chosen by the laboring woman.
  The researcher, wearing gloves, will insert one or two fingers (index and middle) into the participant's vaginal canal and move them from side to side in a "U"-shaped motion, for approximately one second in each direction. Light downward pressure will be applied toward the rectum, according to the woman's tolerance, until relaxation of the massaged perineal muscles is observed.
  A water-based lubricant will be used to facilitate the procedure. The massage will last no longer than 5 minutes.
  Arms: Perineal Massage Group

SUMMARY:
The purpose of this study is to evaluate whether perineal massage during labor can help prevent perineal trauma, such as lacerations or episiotomies.

The study will test two hypotheses:

Null hypothesis: Perineal massage during labor does not prevent perineal trauma.

Alternative hypothesis: Perineal massage during labor helps prevent perineal trauma.

Participants will be randomly assigned to one of two groups:

Perineal massage group: Participants will receive perineal massage during labor.

Control group: Participants will receive the standard care provided by the labor and delivery unit.

A randomization process will be used to assign participants to each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently in labor
* Gestational age between 37 and 42 weeks
* Fetus presenting in cephalic position
* No prior perineal massage performed during prenatal care

Exclusion Criteria:

* Patients who progress to cesarean delivery
* Diagnosis of HELLP syndrome
* Unstable vital signs of the laboring woman or fetus

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 466 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of perineal trauma (laceration or episiotomy) during vaginal delivery | At the time of delivery
  The presence and degree of perineal trauma will be assessed after delivery by the attending healthcare provider. Trauma will be classified by the presence of spontaneous perineal lacerations (graded I to IV) and/or performance of episiotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT07099690/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT07099690/ICF_001.pdf